CLINICAL TRIAL: NCT00789555
Title: Safety of PATANASE® Nasal Spray in Patients With Perennial Allergic Rhinitis
Brief Title: Safety of PATANASE Nasal Spray in Patients With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-08-32
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-01

CONDITIONS: Perennial Allergic Rhinitis
Keywords: nasal allergy; nasal spray; seasonal allergy; perennial allergy
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Seasonal | interventions — Olopatadine Hydrochloride; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PATANASE (Experimental): Olopatadine hydrochloride 0.6% nasal spray (PATANASE), two sprays in each nostril twice a day (morning and evening) for up to 12 months
  Interventions: Drug: Olopatadine hydrochloride 0.6% nasal spray (PATANASE)
- Patanase Vehicle, pH 3.7 (Placebo Comparator): Olopatadine nasal spray vehicle, pH 3.7, two sprays in each nostril twice a day (morning and evening) for up to 12 months
  Interventions: Other: Olopatadine nasal spray vehicle, pH 3.7
- Patanase Vehicle, pH 7.0 (Placebo Comparator): Olopatadine nasal spray vehicle, pH 7.0, two sprays in each nostril twice a day (morning and evening) for up to 12 months
  Interventions: Other: Olopatadine nasal spray vehicle, pH 7.0

INTERVENTIONS:
Drug: Olopatadine hydrochloride 0.6% nasal spray (PATANASE) — Two sprays in each nostril twice a day (morning and evening) for up to 12 months
  Other Names: PATANASE®
  Arms: PATANASE
Other: Olopatadine nasal spray vehicle, pH 3.7 — Two sprays in each nostril twice a day (morning and evening) for up to 12 months
  Arms: Patanase Vehicle, pH 3.7
Other: Olopatadine nasal spray vehicle, pH 7.0 — Two sprays in each nostril twice a day (morning and evening) for up to 12 months
  Arms: Patanase Vehicle, pH 7.0

SUMMARY:
The purpose of this study was to assess local nasal adverse effects, as well as systemic effects, of PATANASE nasal spray when compared with Patanase Vehicle, pH 3.7 and Patanase Vehicle, pH 7.0 in patients with perennial allergic rhinitis (PAR).

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent;
2. Normal nasal exam;
3. History of perennial allergic rhinitis;
4. Allergy to perennial allergen documented by allergy testing;
5. Age 12 years and older;
6. Must follow instructions;
7. Must make required study visits;
8. Negative pregnancy test and adequate birth control methods for females of childbearing potential;
9. Refrain from certain allergy medications during the study;
10. Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

1. Nasal disorders;
2. Use of substances that affect the nasal septum;
3. Exposure to industrial metal plating solutions;
4. Uncontrolled, severe, or unstable diseases;
5. Hypersensitivity to the study drug or nasal spray components;
6. Relative of site staff with access to the protocol;
7. Participation in another investigational study within 30 days or at the same time as this study;
8. Medical Monitor decision;
9. Other protocol-defined exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1260 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center For Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited and enrolled from 69 US study centers.
Pre-assignment Details: 234 subjects were enrolled under protocol Version 1.0, then exited due to a revision in the study plan. A new cohort of 1026 subjects was enrolled in protocol Version 2.0, for a total enrollment of 1260 subjects.
Groups:
- PATANASE; Patanase Vehicle, pH 3.7; Patanase Vehicle, pH 7.0: Two sprays in each nostril twice a day for up to 12 months
Period: Overall Study
Arm/Group | PATANASE | Patanase Vehicle, pH 3.7 | Patanase Vehicle, pH 7.0
Started | 421 | 417 | 422
Completed | 262 | 278 | 263
Not Completed | 159 | 139 | 159
Not completed — Protocol Amendment | 78 | 76 | 80
Not completed — Adverse Event | 17 | 7 | 10
Not completed — Lost to Follow-up | 9 | 10 | 18
Not completed — Patient decision unnrelated to adv event | 38 | 29 | 26
Not completed — Treatment failure | 11 | 8 | 12
Not completed — Protocol Violation | 6 | 9 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PATANASE | Patanase Vehicle, pH 3.7 | Patanase Vehicle, pH 7.0 | Total
Number analyzed (Participants) | 421 | 417 | 422 | 1260
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (14.5) | 36.2 (14.2) | 38.3 (14.6) | 37.1 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 260 | 278 | 789
  Male | 170 | 157 | 144 | 471
Region of Enrollment [Number; unit: participants]
  United States | 421 | 417 | 422 | 1260

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Clinically Relevant Change From Baseline (Day 0) in Nasal Examination Parameters to Exit (Month 12 or Sooner)
Description: Percentage of subjects with clinically relevant change from baseline in protocol-specific safety parameters to time of exit, based on the assessment of the investigator, regardless of causality (related or not related) to test article.
Time Frame: Baseline (Day 0), Exit (Month 12 or sooner)
Population: This analysis population includes all subjects who received study drug (Safety Analysis Set), minus any missing data.
Measure: Number; unit: Percentage of subjects
Arm/Group | PATANASE | Patanase Vehicle, pH 3.7 | Patanase Vehicle, pH 7.0
Number analyzed (Participants) | 386 | 386 | 381
Percentage of subjects
  Anatomic Abnormalities | 0.8 | 1.3 | 0.3
  Bleeding | 0.8 | 1.0 | 2.6
  Infection | 0.3 | 1.0 | 0.0
  Possible Ulcerations | 0.5 | 0.5 | 1.6

2. Secondary Outcome: Percentage of Subjects With Change From Baseline (Day 0) in Pulse Rate Beats Per Minute (BPM) to Exit (Month 12 or Sooner)
Description: Percentage of subjects with change from baseline in pulse measurement to time of exit, as recorded based on a full 60-second count after the patient rested for five minutes.
Time Frame: Baseline (Day 0), Exit (Month 12 or sooner)
Population: Safety Analysis Set, minus any missing data.
Measure: Number; unit: Percentage of subjects
Arm/Group | PATANASE | Patanase Vehicle, pH 3.7 | Patanase Vehicle, pH 7.0
Number analyzed (Participants) | 416 | 414 | 418
Percentage of subjects
  Decrease greater than 30 BPM | 0.0 | 0.0 | 0.0
  Decrease 21-30 BPM | 0.7 | 1.2 | 0.5
  Decrease 11-20 BPM | 7.5 | 9.2 | 6.2
  Decrease 1-10 BPM | 27.2 | 30.4 | 34.7
  No Change | 7.5 | 6.5 | 7.9
  Increase 1-10 BPM | 38.7 | 38.9 | 39.7
  Increase 11-20 BPM | 16.8 | 9.9 | 8.9
  Increase 21-30 BPM | 1.4 | 3.6 | 1.4
  Increase greater than 30 BPM | 0.2 | 0.2 | 0.7

3. Secondary Outcome: Percentage of Subjects With Change From Baseline (Day 0) in Blood Pressure (Systolic) to Exit (Month 12 or Sooner)
Description: Percentage of subjects with change from baseline in systolic blood pressure to time of exit, as obtained in a sitting position after the subject rested for five minutes. Two measurements, separated by two minutes, were obtained, from which the average systolic pressure was derived. If the first two readings differed by more than 5 millimeters of mercury (mmHg), a third reading was taken two minutes later and all three were used to determine the average. The first appearance of sound (phase 1) was used to define systolic blood pressure.
Time Frame: Baseline (Day 0), Exit (Month 12 or sooner)
Population: Safety Analysis Set, minus any missing data.
Measure: Number; unit: Percentage of subjects
Arm/Group | PATANASE | Patanase Vehicle, pH 3.7 | Patanase Vehicle, pH 7.0
Number analyzed (Participants) | 416 | 413 | 418
Percentage of subjects
  Decrease greater than 30 mmHg | 0.5 | 1.2 | 0.5
  Decrease 21-30 mmHg | 1.0 | 2.4 | 2.4
  Decrease 11-20 mmHg | 11.8 | 9.2 | 10.0
  Decrease 1-10 mmHg | 35.3 | 36.3 | 35.4
  No change | 4.6 | 5.3 | 5.3
  Increase 1-10 mmHg | 35.1 | 33.4 | 34.4
  Increase 11-20 mmHg | 10.6 | 10.2 | 10.5
  Increase 21-30 mmHg | 1.2 | 1.9 | 1.2
  Increase greater than 30 mmHg | 0.0 | 0.0 | 0.2

4. Secondary Outcome: Percentage of Subjects With Change From Baseline (Day 0) in Blood Pressure (Diastolic) to Exit (Month 12 or Sooner)
Description: Percentage of subjects with change from baseline in diastolic blood pressure to time of exit, as obtained in a sitting position after the subject rested for five minutes. Two measurements, separated by two minutes, were obtained, from which the average systolic pressure was derived. If the first two readings differed by more than 5 millimeters of mercury (mmHg), a third reading was taken two minutes later and all three were used to determine the average. The disappearance of sound (phase 5) was used to define diastolic blood pressure.
Time Frame: Baseline (Day 0), Exit (Month 12 or sooner)
Population: Safety Analysis Set, minus any missing data.
Measure: Number; unit: Percentage of subjects
Arm/Group | PATANASE | Patanase Vehicle, pH 3.7 | Patanase Vehicle, pH 7.0
Number analyzed (Participants) | 416 | 413 | 418
Percentage of subjects
  Decrease greater than 30 mmHg | 0.0 | 0.2 | 0.2
  Decrease 21-30 mmHg | 0.7 | 1.0 | 0.5
  Decrease 11-20 mmHg | 8.7 | 13.6 | 11.5
  Decrease 1-10 mmHg | 44.5 | 38.7 | 42.6
  No change | 7.5 | 6.1 | 6.5
  Increase 1-10 mmHg | 33.2 | 33.4 | 33.7
  Increase 11-20 mmHg | 5.3 | 6.5 | 5.0
  Increase 21-30 mmHg | 0.2 | 0.5 | 0.0
  Increase greater than 30 mmHg | 0.0 | 0.0 | 0.0

5. Secondary Outcome: Percentage of Subjects With Clinically Relevant Change From Baseline (Day 0) in Physical Examination Parameters to Exit (Month 12 or Sooner)
Description: as for outcome 1
Time Frame: Baseline (Day 0), Exit (Month 12 or sooner)
Population: Safety Analysis Set, minus any missing data.
Measure: Number; unit: Percentage of subjects
Arm/Group | PATANASE | Patanase Vehicle, pH 3.7 | Patanase Vehicle, pH 7.0
Number analyzed (Participants) | 404 | 403 | 392
Percentage of subjects
  Head/EENT | 5.2 | 4.2 | 4.6
  Neck | 0.0 | 0.7 | 0.0
  Cardiovascular | 0.0 | 0.5 | 0.3
  Pulmonary | 0.7 | 0.2 | 0.3
  Abdomen | 0.0 | 0.0 | 0.3
  Skin and Extremities | 1.2 | 0.5 | 1.3
  Neurological | 0.7 | 0.0 | 0.0
  Lymph Nodes | 0.0 | 0.2 | 0.0
  Musculoskeletal | 0.0 | 0.5 | 0.5

6. Primary Outcome: Self-Rated Relief Assessment at Day 30
Description: Relief assessment as rated by the subject on a 4-point scale, where 1=complete relief and 4=no relief. The subject answered the following question: "I would rate the study medication's effectiveness for relieving my allergy symptoms since my last visit as: (1) Complete Relief; (2) Moderate Relief; (3) Mild Relief; (4) No Relief."
Time Frame: Day 30
Population: Analysis population included all subjects enrolled under protocol Version 2.0 who received study drug and attended at least one on-therapy study visit (ITT). The LOCF (last observation carried forward method) was used to impute missing data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PATANASE | Patanase Vehicle, pH 3.7 | Patanase Vehicle, pH 7.0
Number analyzed (Participants) | 328 | 331 | 330
Units on a scale | 2.4 (0.9) | 2.7 (1.0) | 2.7 (0.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 2 years, 1 month, 16 days. Adverse events were defined as any untoward (unfavorable and unintended) medical occurrence in a subject administered a test article.
Description: Adverse events were collected after the first dose of study medication at Visit 1 and during each monthly on-therapy study visit through Visit 13 (or Early Exit). Safety Analysis Set was used for analysis.
Arm/Group | PATANASE | Patanase Vehicle, pH 3.7 | Patanase Vehicle, pH 7.0
Serious Adverse Events (participants affected / at risk) | 8/421 | 7/417 | 14/422
Other Adverse Events (participants affected / at risk) | 220/421 | 213/417 | 214/422
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PATANASE (N=421) | Patanase Vehicle, pH 3.7 (N=417) | Patanase Vehicle, pH 7.0 (N=422)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — Not related
Anxiety (Psychiatric disorders) | 0 | 0 | 1 — Not related
Appendicitis (Infections and infestations) | 0 | 1 | 1 — Not related
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 — Not related
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 1 — Not related
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 — Not related
Cellulitis (Infections and infestations) | 0 | 0 | 1 — Not related
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 1 — Not related
Chest Pain (General disorders) | 1 | 0 | 1 — Not related
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 — Not related
Cystostomy closure (Surgical and medical procedures) | 1 | 0 | 0 — Not related
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 — Not related
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0 — Not related
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 — Not related
Herpes zoster oticus (Infections and infestations) | 0 | 0 | 1 — Not related
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0 — Not related
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0 — Not related
Injury (Injury, poisoning and procedural complications) | 1 | 1 | 1 — Not related
Internal fixation of fracture (Surgical and medical procedures) | 1 | 0 | 0 — Not related
Intravertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Not related
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 — Not related
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 — Not related
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1 — Not related
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 — Not related
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Not related
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 — Related
Sialoadenitis (Infections and infestations) | 1 | 0 | 0 — Not related
Spinal fusion surgery (Surgical and medical procedures) | 0 | 0 | 1 — Not related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PATANASE (N=421) | Patanase Vehicle, pH 3.7 (N=417) | Patanase Vehicle, pH 7.0 (N=422)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 92 | 76 | 85
Headache (Nervous system disorders) | 24 | 27 | 25
Injury (Injury, poisoning and procedural complications) | 31 | 28 | 37
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 31 | 27 | 35
Nasopharyngitis (Infections and infestations) | 50 | 51 | 48
Rhinitis (Infections and infestations) | 51 | 59 | 61
Sinusitis (Infections and infestations) | 55 | 48 | 49
Upper respiratory tract infection (Infections and infestations) | 36 | 52 | 45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right of prior review of any publication or presentation of information related to the study.